CLINICAL TRIAL: NCT06435247
Title: The Effect of Accompaniment by Older Adults on Anaesthetic Recovery
Brief Title: The Effect of Accompaniment by Older Adults on Anesthetic Recovery
Acronym: AAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American British Cowdray Medical Center (Other)
Responsible Party: Principal Investigator, Mariana Guadalupe García Hernandez, Physician investigator, American British Cowdray Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CMABC-24-18
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-07

CONDITIONS: Elderly; Anesthesia; Reaction
Keywords: ancianos; añadir la calidad de la recuperación anestésica; añadir acompañamiento

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial design with two groups
  * One group will have family accompaniment in the recovery area, the other will not
  * The QoR-15 scale will be used to measure the quality of anesthetic recovery
  * The randomization was done using the OpenEpi software
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accompaniment in the recovery area (Experimental): The first group will have a family member accompany them in the recovery area
  Interventions: Behavioral: With or without accompaniment in the recovery anaesthetic area
- without accompaniment (No Intervention): The second group will not have accompaniment as is currently standard practice

INTERVENTIONS:
Behavioral: With or without accompaniment in the recovery anaesthetic area — one grup will have family accompaniment in the recovery area and the other group will not in both groups the QoR15 scale will be used to measure the quality of anesthetic recovery
  Arms: Accompaniment in the recovery area

SUMMARY:
Summary:

In 2022, Mexico estimated a population of 17,958,707 older adults. With increased life expectancy, it is essential to seek strategies that improve the health of this population, as they are more vulnerable compared to other age groups due to functional and cognitive decline, along with an increase in chronic diseases and medication intake. During this stage of life, there is a possibility of requiring surgical treatment, which is the focus of this protocol proposing a maneuver that impacts patients' health without requiring economic costs. The proposal suggests the accompaniment of older adults by a family member during the immediate post-anesthetic period. Hypothesis: Accompaniment of older adults during the immediate postoperative period improves the quality of anesthetic recovery by 60%. This value is based on a study by Shem, where accompanying older adults prior to anesthetic induction resulted in a 61% reduction in anxiety among older adults. Anesthesiologists have expanded their role in perioperative medicine alongside geriatric medicine services for older surgical patients.

An experimental study will be conducted with two randomly divided groups: one group with accompaniment and one group without accompaniment in the recovery area. Both groups will be assessed using different questionnaires: 1. Pfeiffer Test for cognitive impairment diagnosis, 2. QoR-15 to assess the quality of anesthetic recovery, 3. Beck Anxiety Questionnaire, all of which will be administered 24 hours after surgery. Delirium will also be assessed using NuDESC at 24 hours, day 5, and 30 days after surgery. General data prior to surgery will be recorded, and vital signs such as heart rate, blood pressure, and pain on a verbal scale from 0 to 10 will be monitored during the postoperative period.

Statistical analysis will involve representing baseline characteristics of the population using mean and standard deviation or median and interquartile range, depending on the distribution type. X2 will be used to compare both groups in terms of outcomes. Finally, a multivariate analysis will be conducted using logistic regression to adjust for confounding variables.

DETAILED DESCRIPTION:
Justification:

Due to the increase in life expectancy and the growing number of older adults worldwide and in our country, it is important to search for and implement feasible and cost-free measures to improve the quality of medical care, specifically in surgical treatments that impact the reduction of complications, shorten recovery time, and indirectly improve the quality of life for these patients.

Feasibility and relevance:

* The research question aims to improve the quality of medical care for older adults with a humanistic approach.
* In a group of people that will continue to grow, with a longer life expectancy, they will require surgical treatments.
* There are no articles evaluating the quality of anesthetic recovery or its impact on their health with accompaniment.
* Approximately 222 surgeries are performed in this population every month, making it a frequent occurrence.
* It is a measure that does not incur any cost.
* It can be applied in any hospital setting.

Problem statement:

The increase in life expectancy worldwide has led to a larger population of older adults, and Mexico is no exception. Therefore, it is important to establish measures that improve the quality of medical care and reduce complications in this age group, using measures that do not incur any economic costs. Specifically, in the perioperative period, proposing the accompaniment of older adults in the anesthetic recovery area.

Research question:

Does the accompaniment of older adults improve the quality of anesthetic recovery with a score higher than 122 on the QoR15 (quality of recovery - 15) scale?

Hypotheses:

Null hypothesis:

The accompaniment of older adults in the immediate postoperative period does not improve the quality of anesthetic recovery with a score lower than 121 on the QoR15 scale.

Alternative hypothesis:

The accompaniment of older adults in the immediate postoperative period improves the quality of anesthetic recovery with a score higher than 122 on the QoR15 scale.

Overall objective:

- Determine if the accompaniment of older adults improves the quality of anesthetic recovery, classified as good or excellent according to the QoR15 scale with a score of 122 to 150.

Specific objectives:

* Determine the incidence of anxiety in older adults in the anesthetic recovery area, considering anxiety with a score higher than 22 on the Beck scale.
* Determine the presence or absence of delirium in older adults in the perioperative period.
* Assess if the accompaniment of older adults reduces the length of stay in the anesthetic recovery area, aiming for a stay of no more than 60 minutes.

ELIGIBILITY:
Inclusion Criteria: Scheduled for elective surgery under balanced anesthesia with a hospital stay not exceeding 48 hours.

* ASA (American society of anesthesiologist) I y II
* Education level Hight school or higher

Exclusion Criteria:

* History of diseasses associated with dementia
* Emergency surgery.
* Regional anesthesia or sedation
* Moderate to severe cognitive impairment
* History of smoking or drugs
* Surgerios with risk of major bleeding more or equal 1000ml
* Hip or long bone surgeries

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The best score in the QoR15 (Quality of recovery-15) scale greater than 122 | Within 24 hours followin the surgical procedure
  The goal is to evaluate the impact of this accompainment on enhancing the quality of patients anesthetic recovery, as measured by the QoR15 scale

SECONDARY OUTCOMES:
Anxiety in both groups measured using the Beck Anxiety Scale | Before the surgical procedure and 24 hors after the surgical event
  Anxiety will be measured in both groups: the intervetion grup and the control grup. This assessment will occur at two time points
Delirium | 24 hours, day 5 and day 30.
  Delirium will be measured in the two grups at 3 times points post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Garcia, investigator, Principal Investigator — American British Cowdray Medical Center
Locations (2):
- Mexico (2):
  - El Centro Médico American Brithish Cowdray, I.A.P, Mexico City
  - Centro Médico ABC, Mexico City